CLINICAL TRIAL: NCT01422226
Title: IUD Insertion in Nulliparous Women: A Randomized, Placebo-Controlled Trial of Misoprostol for Cervical Priming
Brief Title: Intra Uterine Device Insertion in Nulliparous Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit participants
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-1060
Record Dates: First submitted 2011-08-22; First posted 2011-08-23 (Estimated); Results first posted 2015-02-26 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-12

CONDITIONS: Contraception
Keywords: IUD; contraception; nulliparous; women
MeSH Terms: interventions — Misoprostol; Alprostadil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental active comparator (Experimental): Drug: Misoprostol
  Experimental: 400 mcg taken sublingually 2 hours prior to IUD insertion
  Interventions: Drug: Misoprostol
- Placebo comparator (Placebo Comparator): Other: Placebo
  Pill identical to study drug in appearance, taste, smell. Taken sublingually 2 hours prior to IUD insertion
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Misoprostol — Experimental: 400 mcg taken sublingually 2 hours prior to IUD insertion
  Other Names: synthetic prostaglandin E1 (PGE1) analog
  Arms: Experimental active comparator
Other: Placebo — Pill identical to study drug in appearance, taste, smell. Taken sublingually 2 hours prior to IUD insertion
  Arms: Placebo comparator

SUMMARY:
Over the last several years, more and more women are choosing intrauterine contraception (IUDs) to meet their birth control needs. The effectiveness of IUDs is very similar to tubal sterilization, with an overall unintended pregnancy rate of less than 1% in the first year, and lower failure rates in subsequent years. Intrauterine contraception has many attributes besides its effectiveness; it is easily reversible, has a low side-effect profile, and provides a long-term solution for contraception (10 years for the copper T380 and 5 years for the levonorgestrel IUD). In addition, using an IUD for birth control requires little on-going effort by the woman to be effective and offers immediate return to fertility with its removal.

The biggest increase in users is among nulliparous women (women who have not had children), due to increased awareness of the safety of modern IUDs in this population, and the many benefits of the method. In fact, The copper IUD (Paragard) is now FDA approved for use in nulliparous women, and the American College of Obstetricians and Gynecologists supports the use of both copper and levonorgestrel IUDs in nulliparous women. The cervix of a nulliparous woman has a smaller diameter which can lead to more difficult and uncomfortable IUD insertions. Many providers avoid offering IUDs to nulliparas because of fears that the procedure will be more difficult, and may require cervical dilation, placement of a paracervical nerve block, or placement under ultrasound guidance, none of which are standard for parous women. The medication misoprostol is a prostaglandin E1 analog. Because of misoprostol's known ability to cause cervical dilation, some family planning providers give their nulliparous patients a dose of this drug prior to IUD insertion. Misoprostol is commonly used to dilate the cervix for similar procedures as in first trimester abortions, hysteroscopy and endometrial biopsies. Its efficacy in cervical priming for IUD insertion is unknown, and some concern exists that uterine contractions caused by the drug may lead to device expulsion or displacement.

In this study, the investigators propose to ask nulliparous women who have undergone contraceptive counseling and decided to use an IUD for birth control to be randomized to the use of misoprostol or placebo prior to their scheduled IUD placement.

DETAILED DESCRIPTION:
Hypothesis: The prostaglandin E1 analog misoprostol will ease insertion of intrauterine contraceptive devices in nulliparous women.

Specific Aim 1: To evaluate the ability to place an IUD in the standard fashion, without ancillary measures, in nulliparous women who have received misoprostol versus placebo Specific Aim 2: To evaluate in nulliparous women who have chosen to receive an IUD whether pre-procedure misoprostol eases pain, compared to placebo Specific Aim 3: To evaluate whether misoprostol reduces the rate of complications of IUD placement, compared to placebo Study drug (misoprostol) is being obtained from the University of Utah Health Sciences Center, which is the main study site. The University of Utah Health Sciences Center has obtained an Investigational New Drug (IND) exemption from the FDA in order to use misoprostol for this use in this study. This study is part of a prospective meta-analysis. Deidentified data will be provided to the other sites in a password protected spreadsheet and sent via encrypted, secure email. No identifiable data will be shared with other sites or via the internet. We did not complete attachment G, use of the internet, because this research is not being done via the internet, and no identifiable data will be accessible via the internet or shared with other sites involved in the study. Only deidentified data will be made available to the other sites involved in the prospective meta-analysis.

ELIGIBILITY:
Inclusion Criteria:

* Desires IUD placement
* 18 years old or older
* negative pregnancy test
* no prior pregnancies beyond 14 6/7 weeks
* no pelvic inflammatory disease (PID) in last 3 months
* no current cervicitis
* no contraindications to IUD insertion (see exclusion criteria below)
* willing to follow-up in 6-8 weeks for a standard IUD follow-up visit
* Determined by her clinician to be an appropriate candidate for an IUD.

Exclusion Criteria:

* Active cervical infection
* current pregnancy
* prior pregnancy beyond 15 weeks' gestation
* uterine anomaly
* fibroid uterus
* copper allergy/Wilson's disease (for Paragard)
* undiagnosed abnormal uterine bleeding
* cervical or uterine cancer
* allergy to misoprostol (study drug)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Teal, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hopspital, The Children's Hospital, Aurora, Colorado, United States

REFERENCES:
- [Background] Ghersi D. Prospective Meta-Analysis Methods Group. The Cochrane Collaboration 2002 [cited July 2, 2008]; Available from: http://www.cochrane.org/docs/pma.htm
- [Background] Saav I, Aronsson A, Marions L, Stephansson O, Gemzell-Danielsson K. Cervical priming with sublingual misoprostol prior to insertion of an intrauterine device in nulliparous women: a randomized controlled trial. Hum Reprod. 2007 Oct;22(10):2647-52. doi: 10.1093/humrep/dem244. Epub 2007 Jul 25. PMID 17652452
- [Background] Crane JM, Healey S. Use of misoprostol before hysteroscopy: a systematic review. J Obstet Gynaecol Can. 2006 May;28(5):373-9. doi: 10.1016/s1701-2163(16)32150-8. PMID 16768880
- [Background] Carbonell JL, Velazco A, Rodriguez Y, Tanda R, Sanchez C, Barambio S, Valera L, Chami S, Valero F, Aragon S, Mari J. Oral versus vaginal misoprostol for cervical priming in first-trimester abortion: a randomized trial. Eur J Contracept Reprod Health Care. 2001 Sep;6(3):134-40. PMID 11763976
- [Background] Tang OS, Ho PC. The pharmacokinetics and different regimens of misoprostol in early first-trimester medical abortion. Contraception. 2006 Jul;74(1):26-30. doi: 10.1016/j.contraception.2006.03.005. Epub 2006 Apr 27. PMID 16781256
- [Background] Allen RH, Goldberg AB; Board of Society of Family Planning. Cervical dilation before first-trimester surgical abortion (<14 weeks' gestation). SFP Guideline 20071. Contraception. 2007 Aug;76(2):139-56. doi: 10.1016/j.contraception.2007.05.001. Epub 2007 Jul 10. PMID 17656184
- [Background] American College of Obstetricians and Gynecologists. ACOG Committee Opinion No. 392, December 2007. Intrauterine device and adolescents. Obstet Gynecol. 2007 Dec;110(6):1493-5. doi: 10.1097/01.AOG.0000291575.93944.1a. PMID 18055754
- [Background] ACOG Committee on Practice Bulletins-Gynecology. ACOG practice bulletin. Clinical management guidelines for obstetrician-gynecologists. Number 59, January 2005. Intrauterine device. Obstet Gynecol. 2005 Jan;105(1):223-32. doi: 10.1097/00006250-200501000-00060. No abstract available. PMID 15625179
- [Background] Trussell J. Contraceptive failure in the United States. Contraception. 2004 Aug;70(2):89-96. doi: 10.1016/j.contraception.2004.03.009. PMID 15288211

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Active Comparator | Placebo Comparator
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Active Comparator | Placebo Comparator | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Ease of IUD Insertion (Use of Ancillary Measures)
Description: The primary outcome is the proportion in each group able to have the IUD inserted in a standard fashion without the ancillary measures of mechanical dilation of the cervix, placement of paracervical nerve block, or using abdominal ultrasound for guidance. The null hypothesis for the primary outcome is that misoprostol does not influence difficulty of insertion.
Time Frame: During the IUD insertion procedure, up to 2 hours
Measure: Number; unit: participants
Arm/Group | Experimental Active Comparator | Placebo Comparator
Number analyzed (Participants) | 1 | 2
participants | 1 | 2

ADVERSE EVENTS:
Arm/Group | Experimental Active Comparator | Placebo Comparator
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No